CLINICAL TRIAL: NCT05225649
Title: Pilot Randomized Controlled Trial to Reduce Obesity Risk Factors During the First 1,000 Days
Brief Title: Health e-Baby: Trial to Reduce Obesity Risk Factors During the First 1,000 Days
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AAAT7915
Record Dates: First submitted 2022-01-17; First posted 2022-02-04 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Obesity, Infant
Keywords: First 1,000 days; Mobile Health; Behavior Change Intervention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be identified by a participant code to the care provider, investigator, and outcomes assessor until primary analysis is complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavior Change Intervention (Experimental): Participants will receive health coaching, patient-directed behavior change support by mobile health, and usual clinical care.
  Interventions: Behavioral: Behavior Change Intervention
- Control (No Intervention): Participants will receive usual clinical care.

INTERVENTIONS:
Behavioral: Behavior Change Intervention — Health coaching sessions; self-monitoring: Fitbit, home scale, and app; personalized health information by mobile health: growth charts and age-specific health behavior information via text message and email; behavior change support by mobile health: family-based health behavior goal setting via chatbot; and usual clinical care.
  Arms: Behavior Change Intervention

SUMMARY:
Specific Aim: Feasibility of a Pilot Randomized Controlled Trial (RCT) in Pregnancy and Infancy to Reduce Childhood Obesity Risk Factors in Early Life.

The main outcomes are feasibility of the intervention components and data collection. Study will use maternal body mass index (BMI) and child weight-for-length outcomes to estimate sample size needed for a full-scale trial to test intervention efficacy. Primary analysis for full-scale trial power and sample size calculations will be conducted using child weight-for-length data at Child Age 12 Months Visit. Data collected will inform future interventions.

DETAILED DESCRIPTION:
Early life interventions to prevent childhood obesity among disproportionately burdened populations are needed to reduce childhood obesity.

The overall goal of this study is to test the feasibility of a pilot randomized controlled trial to promote healthy maternal weight in pregnancy and post-partum and normal child weight-for-length from birth to age 12 months. The study will include 50 women (enrollment up to 70 to account for potential attrition) in pregnancy and their child through age 12 months to examine rates of study component completion, study component satisfaction, and retention. Women enrolled in the intervention will participate in virtual health coaching and receive self-directed behavior change materials by text and email. The results of this study will help us develop efficacious childhood obesity prevention interventions and determine how many study participants would be needed for a full-scale trial. Ultimately, this research could open new avenues for studying ways to promote health starting early in life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years at time of enrollment
* Gestational age 10-20 weeks at time of enrollment
* Receiving primary care or prenatal care at Columbia/New-York Presbyterian site
* Planned delivery at Columbia/New-York Presbyterian with planned continuation of primary care (postpartum and pediatric) at Columbia/New-York Presbyterian
* Ability to read and respond to questions in English or Spanish
* Smart phone ownership
* Willingness to receive information by smart phone for 18-month intervention and follow-up duration
* Willingness to be randomized into an observational study or an intervention and complete all study components
* Gives permission to participate in receiving messages to their smart phone and email
* Gives permission to complete all study procedures
* Has a physician's clearance for light to moderate physical activity
* Has an active email address
* Capable of providing informed consent
* Has access to Wi-Fi connection in their household

Exclusion Criteria:

* Multiple gestation
* Pre-pregnancy body mass index <18.5 kg/m2 >40
* Major fetal anomaly
* Fetal genetic abnormality
* Planned termination of pregnancy
* Chronic medical conditions that affect nutrition or prohibit regular exercise or alter weight status such as:
* Diseases associated with glucose metabolism
* Diabetes (Type 1, type 2)
* Inflammatory Bowel Disease (Crohn's disease, ulcerative colitis)
* History of gastric bypass/gastric sleeve
* Uncontrolled thyroid disease (hypo or hyperthyroidism)
* Condition requiring enteral tube feeding
* Congenital or acquired heart disease that impacts nutritional needs and physical activity ability
* HIV/AIDS
* Kidney disease
* Cancer
* Uncontrolled autoimmune disease
* Lupus
* Multiple sclerosis
* Sickle cell disease
* Zika infection
* Taking or planning to take certain prescription medications including high dose glucocorticoids, atypical antipsychotics associated with weight gain (such as risperdal (risperidone), clozapine (clozaril), olanzapine (zyprexa), quetiapine (seroquel), etc.), or other prescription weight loss medications
* Personal history of breast cancer or any other type of cancer other than a basal cell skin cancer
* Personal history of cardiovascular disease (coronary artery disease, congestive heart failure, valvular heart disease, stroke, transient ischemic attack, or intermittent claudication), kidney disease, liver disease, venous or arterial thromboembolic disease, adrenal insufficiency, depression requiring hospitalization within the past 6 months, or non-pregnancy related illness requiring overnight hospitalization in the past 6 months
* Underlying disease/treatment that might interfere with participation in/completion of the study (e.g., significant gastrointestinal conditions, major psychiatric disorders, and others at the discretion of the study clinician)
* Other active medical problems detected by examination or laboratory testing
* Inability to complete study visits or intervention components
* Unwillingness or inability to commit to a 18-month research study for them or their child, including plans to move away
* Plans to be in a different geographic area within the next 2 years
* Unable to give informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Arm specific retention rates at 18 months | Up to 18 months
  The retention rate will be defined as the proportion of enrolled individuals who complete infant age 12-months study visits (study month 18) according to each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Mencin, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No